CLINICAL TRIAL: NCT00001650
Title: Studies of Lymphocyte Kinetics Using Bromodeoxyuridine
Brief Title: Use of Bromodeoxyuridine to Study White Blood Cell Replication and Survival in HIV-Infected Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970189; 97-I-0189
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-13

CONDITIONS: HIV Infection; Acquired Immunodeficiency Syndrome
Keywords: BrDU; HIV; Labeling; CD4 Cells; Immunodeficiency
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Immunologic Deficiency Syndromes

SUMMARY:
This study will examine how quickly white blood cells called CD4 lymphocytes reproduce and how long they live in people infected with HIV. It will do this using bromodeoxyuridine (BrDU), a compound that is structurally similar to thymidine, one of the building blocks of DNA. BrDU gets incorporated into DNA instead of thymidine, but it can only get into cells that are replicating. Therefore, measuring the proportion of cells with BrDU indicates how many cells are replicating.

HIV-infected patients 18 years of age and older may be eligible for this study. Candidates will be screened with a medical history, physical examination, chest X-ray, electrocardiogram (EKG) and blood tests.

Participants will be given an infusion of BrDU through a catheter (thin plastic tube) placed in an arm vein. Blood will be drawn up to 4 times in the first 24 hours after the infusion.

Additional samples will then be collected as often as daily for the first week, twice a week for the next 3 weeks and then weekly to monthly for up to 1 year. Some patients may undergo a tissue biopsy (removal of a small tissue sample from a lymph node, tonsil or colon) or computed tomography (CT) scans of the thymus (a small gland between the lungs that manufactures lymphocytes. Some patients will have a second infusion in order to examine changes in the rate of CD4 replication over time or following potent antiretroviral therapy. Patients will be followed in the clinic periodically for the first year and then will be seen in the clinic or contacted by telephone once a year for 4 more years.

The results of this study may provide a better understanding of how HIV causes disease and how therapy affects the immune system.

DETAILED DESCRIPTION:
Understanding the rate of lymphocyte replication and destruction in HIV infected patients, as well as the effects of therapy on lymphocyte replication should lead to a better understanding of the mechanisms behind the immunodeficiency induced by HIV. To examine this directly, up to 85 HIV-infected patients will be enrolled in the study. Patients will receive up to two 30 minute infusions (at least one month apart) of bromodeoxyuridine (BrDU; 200 mg/m(2)), an analogue of thymidine. BrDU is incorporated into DNA and can be measured using an anti-BrDU monoclonal antibody. It can be measured in subpopulations of cells to determine the rate of replication of those cells. All participants in this study will be reimbursed for the inconvenience and discomfort associated with study participation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  18 years or older.

Documented HIV infection (ELISA/Western blot positive or, for acute seroconverters, PCR positive).

Able to provide informed consent and willing to comply with study requirements and clinic policies.

Negative urine or serum pregnancy test (for women of childbearing potential). In addition, women of childbearing potential must agree to practice abstinence or use two methods of birth control / contraception for 4 weeks prior to and 2 weeks after each BrDU infusion. Similarly, all men must agree to practice abstinence or use a condom when engaging in intercourse during the same time period.

Hemoglobin greater than 9 mg/dl; platelets greater than 50,000/mm(3); neutrophils greater than 750 cells/mm(3).

AST/ALT less than 300 IU/ml.

Less than Grade 2 level toxicity for other laboratory parameters.

EXCLUSION CRITERIA:

Active substance abuse or prior history of substance abuse which may interfere with protocol compliance.

Psychiatric illness or disturbance which, in the assessment of the protocol team, may affect safety or compliance.

Significant underlying cardiac, pulmonary, renal, gastrointestinal, rheumatologic or CNS disease as detectable on routine history, physical exam, or screening laboratory studies.

Pregnancy or breast-feeding.

Ongoing therapy with topical or systemic 5-fluorouracil.

Willingness to allow stored samples to be used for future studies of HIV infections and immunological function, and willingness to have HLA typing performed.

Patients who are virologic responders and immunologic non-responders (10-15 patients):

Plasma HIV less than 500 copies/ml by bDNA or RT-PCR for 1 year while receiving HAART, which includes at a minimum 3 antiretroviral drugs, at least one of which is a protease inhibitor or non-nucleoside reverse transcriptase inhibitor, and plasma HIV less than 50 copies /ml by the bDNA assay, performed at the NIH, within the 4 weeks prior to enrollment;

CD4 count less than 300 cells/mm(3) on 2 occasions at least one week apart, with no documented CD4 count greater than 350 cells/mm(3) during the prior 6 months;

No ongoing opportunistic infection or malignancy.

Patients who are virologic and immunologic responders (10-15 patients, matched if possible to study group for age (+/- 5 years) and duration of HAART therapy (+/- 6 months):

Plasma HIV less than 500 copies/ml by bDNA or RT-PCR for 1 year while receiving HAART, which includes at a minimum 3 antiretroviral drugs, at least one of which is a protease inhibitor or non-nucleoside reverse transcriptase inhibitor, and plasma HIV less than 50 copies/ml by the bDNA assay, performed at the NIH, within the 4 weeks prior to enrollment;

CD4 count greater than 350 cells/mm(3) on 2 occasions at least one week apart; CD4 count prior to the initiation of HAART therapy documented to be less than 300 cells/mm(3);

No ongoing opportunistic infection or malignancy.

For all patients: Willingness to have a CT scan of the thymus, to be performed under protocol 95-I-0027.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 1997-09-19; Study Completion 2011-05-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ho DD, Neumann AU, Perelson AS, Chen W, Leonard JM, Markowitz M. Rapid turnover of plasma virions and CD4 lymphocytes in HIV-1 infection. Nature. 1995 Jan 12;373(6510):123-6. doi: 10.1038/373123a0. PMID 7816094
- [Background] Wolthers KC, Bea G, Wisman A, Otto SA, de Roda Husman AM, Schaft N, de Wolf F, Goudsmit J, Coutinho RA, van der Zee AG, Meyaard L, Miedema F. T cell telomere length in HIV-1 infection: no evidence for increased CD4+ T cell turnover. Science. 1996 Nov 29;274(5292):1543-7. doi: 10.1126/science.274.5292.1543. PMID 8929418
- [Background] Sprent J, Tough DF. Lymphocyte life-span and memory. Science. 1994 Sep 2;265(5177):1395-400. doi: 10.1126/science.8073282.